CLINICAL TRIAL: NCT06856460
Title: The Impact of Low Glycemic Index Nutritional Shake on Glucose Regulation in Overweight and Obese Adults
Acronym: SHAKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Stavros Kavouras, Professor and Assistant Dean, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00016899
Record Dates: First submitted 2025-02-25; First posted 2025-03-04 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Hyperglycemia; Obesity Prevention
Keywords: meal replacement; glucose regulation
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Two arms: one group will undergo 2 weeks of a meal replacement shake for breakfast with oat cereal and the other group will consume only oat cereal (isocaloric 400 kilocarolies)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control: Breakfast with 400 kcal of oat cereal with honey (Sham Comparator)
  Interventions: Dietary Supplement: Ceral Breakfast
- Experimental: Breakfast with 200 kcal of oat ceral with honey + 200 kcal of glucose assist shake. (Experimental)
  Interventions: Dietary Supplement: powder shake with very low glycemic index

INTERVENTIONS:
Dietary Supplement: powder shake with very low glycemic index — 2 weeks of cereal and standard process glucose assist shake as part of breakfast. The diet for the remainder of the day will remain unchanged.
  Arms: Experimental: Breakfast with 200 kcal of oat ceral with honey + 200 kcal of glucose assist shake.
Dietary Supplement: Ceral Breakfast — consume of 400kcal of oat-based cereal with honey for breakfast
  Arms: Control: Breakfast with 400 kcal of oat cereal with honey

SUMMARY:
Low glycemic index nutritional shakes have clinically shown to improve post-prandial glycemic responses in acute laboratory control studies. However, there is limited information on how replacing meals with low-glycemic index shake could impact glucose regulation in free-living adults consuming their own diets.

The present study aims to examine the impact of adding the SP Glucose-Assist shake to the breakfast of non-diabetic overweight and obese adults.

Subjects:

40 non-diabetic adults aged 25-65 years and body mass index ranging between 25-39 .

Protocol:

This is going to be a three-week study that will include a one-week self-selected diet, followed by two weeks of a breakfast supplement shake (standard process glucose assist) or control cereal oat breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 25-40
* Eating pattern 3 meals a day
* stable weight for the last 2 months (<5 pounds fluctuation)
* Willing to eat oat cereal for breakfast
* glycated hemoglobin <7%

Exclusion Criteria:

* glycated hemoglobin >7%
* Body mass index ≤25 or ≥ 40
* Night shifting work
* Atypical meal pattern (not three meals a day or intermittent fasting)
* Thyroid medication
* Bariatric surgery
* Habitual strenuous exercise
* Commuting by bicycle
* Eating disorders
* Use of aspirin during the duration of the study
* Intake of Vit C >60 mg/day during the study
* cancer
* cardiovascular disease
* renal disease
* hepatic disease
* X-ray, MRI or CT appointment during the study duration
* Current infection requiring medication
* Chronic, contagious, infectious diseases such as tuberculosis, Hepatitis A, B, C, or HIV
* Medications of supplements that could affect body weight or appetite (i.e. Ozempic)
* Participating in another study at the same time

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Glucose response between two breakfasts | the entire 2 hours of the glycemic test
  The difference between the two breakfasts on the positive integer of the area under the curve for glucose during the 2 hours following breakfast ingestion.
Insulin responses between the two breakfasts | The entire 2 hours period
  The difference between the two breakfasts on the positive integer of the area under the curve for insulin; during the 2 hours following breakfast ingestion.
Glucose réponses during glucose challenge test | 2 hours post ingestion of the emperimental meal (cereal or ceral + shake)
  Positive integer of the area under the curve for glucose during the 2 hours glycemic test
Insulin responses during the glucemic challenge test | 2 hour post ingestion of the intervention meal (cereal or cereal + shake)
  Positive integer of the area under the curve for insulin during the 2-hours glycemic test

SECONDARY OUTCOMES:
Ambulatory glucose profile | total area under the curve during the 2 weeks (14 days) of dietary intervention.
  The difference between the two groups on the area under the curve in Ambulatory glucose measured with a continuous glucose monitor during the 2 weeks of dietary intervention.
Blood glucagon | 0, 30, 60, 90, and 120 minutes of the glycemic test.
  Blood glucagon difference between day 7 and day 21 during the 2 hours glycemic challenge (400 kilocalories consumption of the oat or oat and glucose assist shake)
Glucagon like peptide 1 | 0, 30, 60, 90, and 120 minutes of the glycemic test.
  Blood Glucagon like peptide difference between day 7 and day 21 during the 2 hours glycemic challenge (400 kilocalories consumption of the oat or oat and glucose assist shake)
Leptin | 0, 30, 60, 90, and 120 minutes of the glycemic test.
  Blood Leptin difference between day 7 and day 21 during the 2 hours glycemic challenge (400 kilocalories consumption of the oat or oat and glucose assist shake)
Adiponectin | 0, 30, 60, 90, and 120 minutes of the glycemic test.
  Blood Adiponectin difference between day 7 and day 21 during the 2 hours glycemic challenge (400 kilocalories consumption of the oat or oat and glucose assist shake)
Ghrelin | 0, 30, 60, 90, and 120 minutes of the glycemic test.
  Blood Ghrelin difference between day 7 and day 21 during the 2 hours glycemic challenge (400 kilocalories consumption of the oat or oat and glucose assist shake)
C-Peptide | 0, 30, 60, 90, and 120 minutes of the glycemic test.
  Blood c-peptide difference between day 7 and day 21 during the 2 hours glycemic challenge (400 kilocalories consumption of the oat or oat and glucose assist shake)

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University 850 PBC, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No